CLINICAL TRIAL: NCT00136292
Title: An Evaluation of the Pharmacokinetics of a Single Dose of Daptomycin (4 mg/kg) in Pediatric Patients Aged Two to Seventeen Years Who Are Concurrently Receiving Standard Antibiotic Therapy for Proven or Suspected Gram-positive Infection
Brief Title: Study of Single Dose Daptomycin in Pediatric Patients With Gram-positive Infection for Which They Are Receiving Standard Antibiotics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 3009-028; DAP-PEDS-05-01 (Other: Cubist Study Number)
Record Dates: First submitted 2005-08-25; First posted 2005-08-29 (Estimated); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Gram-positive Bacterial Infections
Keywords: Gram-Positive Infection
MeSH Terms: conditions — Gram-Positive Bacterial Infections | interventions — Daptomycin

INTERVENTIONS:
Drug: daptomycin

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics of a single dose of daptomycin in patients aged 2-17 years old who have a suspected or proven gram-positive infection for which they are receiving standard antibiotic therapy. The tolerability of a single dose of daptomycin in these patients will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* 2-17 years old
* Suspected or diagnosed gram-positive infection for which the patient is receiving standard antibiotic therapy
* Clinically stable with no evidence of hemodynamic instability in the 72 hour window prior to enrollment, and no history or evidence of renal or hepatic compromise, or clinically significant alterations in fluid/electrolyte homeostasis
* Creatinine clearance (CLcr) ≥ 80 ml/min/1.73 m2 as determined by the Schwartz equation
* Creatine phosphokinase (CPK) levels within normal limits

Exclusion Criteria:

* Known allergy to daptomycin
* History of clinically significant cardiovascular, renal, hepatic, pulmonary (well-controlled asthma is acceptable), gastrointestinal, endocrine, hematologic, or autoimmune disease
* Pneumonia as sole gram-positive infection
* Use of HMG-CoA reductase inhibitors or other systemic anti-hyperlipidemic agents within 7 days prior to study drug administration and expected use through 3 days post-dose
* Clinically significant abnormal laboratory test results (including electrocardiograms [ECGs]), as determined by Investigator
* Body mass index (BMI) that is outside of the 5th to 95th percentile for age
* History (personal or 1st degree relative) of clinically significant muscular disease, nervous system, seizure or psychiatric disorder
* Expected intramuscular (IM) injection within 3 days following dosing
* Expected surgical procedure(s) within 3 days following dosing
* Unexplained muscular weakness
* Rhabdomyolysis, myositis or septic shock

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2005-08-24 (Actual); Primary Completion 2006-08-01 (Actual); Study Completion 2006-08-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic

SECONDARY OUTCOMES:
Tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Richard Jacobs, MD, Principal Investigator — University of Arkansas
Locations (3):
- United States (3):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - University of Texas Southwestern, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Abdel-Rahman SM, Benziger DP, Jacobs RF, Jafri HS, Hong EF, Kearns GL. Single-dose pharmacokinetics of daptomycin in children with suspected or proved gram-positive infections. Pediatr Infect Dis J. 2008 Apr;27(4):330-4. doi: 10.1097/INF.0b013e318160edfc. PMID 18316988